CLINICAL TRIAL: NCT06757036
Title: Effect of Laughter Yoga on Hope and Well-Being Levels of Earthquake Victim Mothers
Brief Title: The Effect of Laughter Yoga on Hope and Well-Being Levels of Earthquake Victim Mothers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Gülcan Bahçecioğlu Turan, Principal Investigator, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ı 2024l13
Record Dates: First submitted 2024-12-27; First posted 2025-01-03 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Laughter Yoga
MeSH Terms: interventions — Laughter Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter Yoga (Experimental): The group where Laughter Yoga is performed
  Interventions: Behavioral: Laughter Yoga
- no Laughter Yoga (No Intervention): he group where Laughter Yoga isn't performed

INTERVENTIONS:
Behavioral: Laughter Yoga — the group where Laughter Yoga is performed
  Arms: Laughter Yoga

SUMMARY:
In Turkey, on February 6, 2023, an earthquake measuring 7.7 in magnitude centered in the Pazarcık district of Kahramanmaraş Province, followed by a second earthquake measuring 7.6 in magnitude centered in Elbistan, caused the deaths of 50,783 people in the provinces of Kahramanmaraş, Gaziantep, Şanlıurfa, Diyarbakır, Adana, Adıyaman, Osmaniye, Hatay, Kilis, Malatya and Elazığ. The magnitude of the cost impact of the 2023 Kahramanmaraş earthquake, which is described as the "disaster of the century" and calculated as 103.6 billion dollars, is as disturbing as the devastating effect of the disaster on individuals' levels of hope and well-being.

In line with previous studies, the high probability that socio-psychological effects will continue for a long time after the February 6, 2023 earthquakes necessitates physical and mental self-care activities to support the health and well-being of those affected by the disaster.

In order for the child's first teacher and guide to be his/her mother and for the widespread impact of our project to reach a wider audience directly and indirectly, the project will address the suitability of laughter yoga as a relaxing practice that will benefit earthquake-stricken mothers living in the provinces of Elazığ and Malatya, which were affected by the 2023 Kahramanmaraş Earthquakes.

Laughter yoga, which has become increasingly popular worldwide and has recently been recognized as a low-cost, risk-free and less time-consuming practice for improving mental health, is a group-based laughter exercise that includes real-life laughter, light movement, stretching, rhythmic breathing and meditation. When articles evaluating the psychological and physiological effects of laughter yoga on individuals are examined, it is observed that promising results are obtained. A recent meta-analysis of 45 interventions that encourage laughter with 2,500 randomized participants found significant positive mental and physical health effects. Although challenging, laughing when sad can be "a great way to balance sadness."

Hope is considered as a situation that includes the individual's high positive expectations for the future, their belief in the world, and the idea that life is worth living. High hope also has a positive effect on coping with traumatic experiences. It is known that individuals' well-being decreases as a result of traumatic life events and that they have difficulty coping with the current situation. In a study conducted on 188 adults who experienced the earthquake that occurred in the Pazarcık and Elbistan districts of Kahramanmaraş on February 6, 2023, it was pointed out that having positive resources such as hope and well-being is important for individuals to cope with post-traumatic symptoms.

Although laughter yoga is expected to support hope and well-being, no study has revealed this relationship after a disaster. Therefore, evidence-based studies are needed to evaluate the effect of laughter yoga on hope and well-being in mothers, who are important building blocks of society after an earthquake. The aim of this study is to clarify the relationship between hope and well-being and laughter yoga after the Kahramanmaraş earthquakes.

ELIGIBILITY:
Inclusion Criteria:

* Having experienced the Kahramanmaraş earthquakes in any of the 11 provinces
* Being willing to participate in the Laughter Yoga practice
* Having a Post-Earthquake Trauma Symptoms Scale score above the threshold value

Exclusion Criteria:

* Those with chronic illnesses that require medical treatment
* Those who report receiving psychiatric treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Post-Earthquake Trauma Symptoms Scale | 3 week
  The scale developed by Tanhan and Kayri (2013) aims to measure trauma symptoms that may occur in individuals after an earthquake. The scale consists of 20 items and 5 dimensions. A score in the range of 52.385±5.051 from the scale corresponds to a threshold value indicating that individuals are traumatized. A value above or below this value indicates high and low levels of showing post-earthquake traumatic symptoms.
Trait Hope Scale: | 3 week
  eveloped by Snyder et al. (1991) and adapted to Turkish by Tarhan and Bacanlı (2015), the scale measures the trait hope levels of individuals aged 15 and over. The scale is an eight-point Likert type and consists of 12 items and two sub-dimensions called Acting Thought and Alternative Paths Thinking. Each of these two sub-dimensions is measured with four items. In this respect, there are also 4 filler items in the scale. These filler items are not scored during scoring. In scoring, only the scores obtained from the Acting Thought and Alternative Paths Thinking sub-dimensions are added up and the total score of these two dimensions is calculated to obtain a total score. The lowest score is 8 and the highest is 64 from the scale.
Psychological Well-Being Scale | 3 week
  The scale, developed by Diener et al. (2009-2010) and adapted to Turkish by Telef (2011; 2013), is a 7-point Likert-type scale that complements existing well-being measurements and does not aim to measure socio-psychological well-being. The lowest score possible from the scale is 8 and the highest is 56. Increasing scores indicate that individuals have many psychological resources and strengths and that their level of psychological well-being is high